CLINICAL TRIAL: NCT05903560
Title: Radial Versus Femoral Access For Thrombectomy in Patients With Acute Basilar Artery Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Xinfeng Liu, Professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RACE-BAO
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the radial group (Experimental): Patients with basilar artery occlusion within 24 hours of onset will be chosen to receive endovascular recanalization via radial approach randomly
  Interventions: Procedure: endovascular recanalization via radial approach
- the femoral group (Active Comparator): Patients with basilar artery occlusion within 24 hours of onset will be chosen to receive endovascular recanalization via femoral approach randomly
  Interventions: Procedure: endovascular recanalization via femoral approach

INTERVENTIONS:
Procedure: endovascular recanalization via radial approach — Patients with basilar artery occlusion within 24 hours of onset will be chosen to receive endovascular recanalization via radial approach
  Arms: the radial group
Procedure: endovascular recanalization via femoral approach — Patients with basilar artery occlusion within 24 hours of onset will be chosen to receive endovascular recanalization via femoral approach
  Arms: the femoral group

SUMMARY:
Stroke is one of the most important diseases endangering the health and quality of life of Chinese people. Acute ischemic stroke (AIS) is commonly caused by cerebrovascular stenosis or occlusion. The most effective treatment for AIS is timely and successful angiographic reperfusion.

Due to the large diameter and obvious positioning of bilateral femoral arteries, the transfemoral artery (TFA) using Seldinger's technique has been the most commonly used approach for endovascular treatment. However, recent studies have suggested that the radial artery is an ideal puncture site for cerebrovascular intervention. Small sample studies have confirmed that endovascular recanalization for acute anterior circulation large vessel occlusion via TRA has been safe and effective. Still, there are some complex approaches needed to be converted to TFA. There has been no difference in total operation duration and fluoroscopy time between TRA and TFA, but the TRA group had higher radiation dose and shorter hospital stays than the TFA group. In addition, TRA tends to be more convenient than TFA, especially for posterior circulation lesions.

However, the current studies are based on a single center with a small sample size, and there has been still a lack of large-sample randomized controlled experiments to verify the safety and effectiveness of posterior endovascular recanalization via TRA.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke in the posterior circulation confirmed by symptoms and imaging examinations.
2. Basilar artery occlusion confirmed by computed tomographic angiography (CTA), magnetic resonance angiography (MRA), or digital subtraction angiography (DSA).
3. Age ≥ 18 years.
4. Time from symptom onset to randomization within 24 hours of the estimated time of basilar artery occlusion.
5. Baseline NIHSS score ≥ 10 before randomization.
6. Intact dual circulation of the hand assessed by the modified Allen's test.
7. Written informed consent from patients or their legally authorized representatives.

Exclusion Criteria:

1. Pre-stroke disability with mRS score ≥ 3.
2. Pregnant or lactating women.
3. Allergic to contrast agents or nitinol devices.
4. Participation in other clinical trials.
5. Systolic blood pressure > 185 mmHg or diastolic blood pressure > 110mmHg, and can not be controlled by antihypertensive drugs.
6. Known genetic or acquired bleeding diathesis, lack of coagulation factors; or oral anticoagulant therapy with INR > 1.7.
7. Baseline lab values: blood glucose < 50mg/dL (2.8mmol/L) or > 400mg/dL (22.2 mmol/L), platelet count < 50*109 /L, or hematocrit < 25%.
8. Life expectancy less than 1 year.
9. Lost to follow-up within 90 days (e.g. no fixed residence, overseas patients, etc.).
10. Acute ischemic stroke within 48 hours after percutaneous coronary intervention, cerebrovascular intervention, or major surgery (patients can be included if more than 48 hours).
11. Clinical manifestations of central nervous system vasculitis.
12. Premorbid nervous system diseases or mental disorders hindering the assessment of the disease.
13. Diseases or anatomical abnormalities that make it difficult for radial or femoral artery puncture, sheath insertion or instrument delivery, such as local infection, anatomical abnormalities confirmed by ultrasound or other imaging examinations, previous interventional or open surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2023-07-22 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
favorable neurological function | at 90 days post-operation
  favorable neurological function (defined as mRS score ≤ 3)

SECONDARY OUTCOMES:
Procedure time | at the operation 1 day
  Procedure time of the endovascular thrombectomy

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, MD, Principal Investigator — Department of Neurology, Jinling Hospital, China
Locations (1):
- Department of Neurology, Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No